CLINICAL TRIAL: NCT06168318
Title: A 3-part, Phase 1, Single-center, Open-label Study to Assess the Relative Bioavailability of Oral Formulations for an Investigational Capsid Inhibitor in Healthy Adult Participants, and to Evaluate the Effect of Food on Bioavailability for an Investigational Capsid Inhibitor in Healthy Adult Participants
Brief Title: A Study to Investigate the Relative Bioavailability and Food Effect of an Oral Capsid Inhibitor Tablet Formulation Compared With Other Oral Tablet Formulations in Male and Female Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 220095
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus; HIV-1; capsid inhibitor; VH4004280; food effect; fasted conditions; fed conditions; bioavailability
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (13):
- Part 1 - Regimen A (Experimental): VH4004280 Formulation A tablet administered in fed conditions.
  Interventions: Drug: VH4004280 Formulation A
- Part 1 - Regimen B (Experimental): VH4004280 Formulation B tablet administered in fed conditions.
  Interventions: Drug: VH4004280 Formulation B
- Part 1 - Regimen C (Experimental): VH4004280 Formulation C tablet administered in fed conditions.
  Interventions: Drug: VH4004280 Formulation C
- Part 1 - Optional Regimen D (Experimental): VH4004280 Formulation D tablet administered in fed conditions.
  Interventions: Drug: VH4004280 Formulation D
- Part 1 - Optional Regimen E (Experimental): VH4004280 Formulation E tablet administered in fed conditions.
  Interventions: Drug: VH4004280 Formulation E
- Part 2 - Regimen A (Experimental): VH4004280 Formulation A tablet administered in fasted conditions.
  Interventions: Drug: VH4004280 Formulation A
- Part 2- Optional Regimen 1 (Experimental): VH4004280 Formulation B, C, D, or E tablet administered in fasted conditions.
  Interventions: Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D; Drug: VH4004280 Formulation E
- Part 2- Optional Regimen 2 (Experimental): VH4004280 Formulation B, C, D, or E tablet administered in fasted conditions.
  Interventions: Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D; Drug: VH4004280 Formulation E
- Part 2- Optional Regimen 3 (Experimental): VH4004280 Formulation B, C, D, or E tablet administered in fasted conditions.
  Interventions: Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D; Drug: VH4004280 Formulation E
- Part 3 - Optional Regimen 1 (Experimental): VH4004280 Formulation A, B, C or D tablet administered in lower fat conditions.
  Interventions: Drug: VH4004280 Formulation A; Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D
- Part 3- Optional Regimen 2 (Experimental): VH4004280 Formulation A, B, C or D tablet administered in lower fat conditions.
  Interventions: Drug: VH4004280 Formulation A; Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D
- Part 3 - Optional Regimen 3 (Experimental): VH4004280 Formulation A, B, C or D tablet administered in lower fat conditions.
  Interventions: Drug: VH4004280 Formulation A; Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D
- Part 3 - Optional Regimen 4 (Experimental): VH4004280 Formulation A, B, C or D tablet administered in lower fat conditions.
  Interventions: Drug: VH4004280 Formulation A; Drug: VH4004280 Formulation B; Drug: VH4004280 Formulation C; Drug: VH4004280 Formulation D

INTERVENTIONS:
Drug: VH4004280 Formulation A — Oral administration of VH4004280 Formulation A in fasted or fed conditions.
  Arms: Part 1 - Regimen A; Part 2 - Regimen A; Part 3 - Optional Regimen 1; Part 3 - Optional Regimen 3; Part 3 - Optional Regimen 4; Part 3- Optional Regimen 2
Drug: VH4004280 Formulation B — Oral administration of VH4004280 Formulation B in fasted or fed conditions.
  Arms: Part 1 - Regimen B; Part 2- Optional Regimen 1; Part 2- Optional Regimen 2; Part 2- Optional Regimen 3; Part 3 - Optional Regimen 1; Part 3 - Optional Regimen 3; Part 3 - Optional Regimen 4; Part 3- Optional Regimen 2
Drug: VH4004280 Formulation C — Oral administration of VH4004280 Formulation C in fasted or fed conditions.
  Arms: Part 1 - Regimen C; Part 2- Optional Regimen 1; Part 2- Optional Regimen 2; Part 2- Optional Regimen 3; Part 3 - Optional Regimen 1; Part 3 - Optional Regimen 3; Part 3 - Optional Regimen 4; Part 3- Optional Regimen 2
Drug: VH4004280 Formulation D — Oral administration of VH4004280 Formulation D in fasted or fed conditions.
  Arms: Part 1 - Optional Regimen D; Part 2- Optional Regimen 1; Part 2- Optional Regimen 2; Part 2- Optional Regimen 3; Part 3 - Optional Regimen 1; Part 3 - Optional Regimen 3; Part 3 - Optional Regimen 4; Part 3- Optional Regimen 2
Drug: VH4004280 Formulation E — Oral administration of VH4004280 Formulation E in fasted or fed conditions.
  Arms: Part 1 - Optional Regimen E; Part 2- Optional Regimen 1; Part 2- Optional Regimen 2; Part 2- Optional Regimen 3

SUMMARY:
This is a 3 part study of an investigational capsid inhibitor, VH4004280, in healthy adult participants. The purpose is to evaluate the effect of tablet formulation as well as food on bioavailability. Part 1 of the study will compare the relative bioavailability of VH4004280 Formulation A tablets to up to 4 alternative tablet formulations under fed (high fat) conditions. Part 2 of the study will assess the effect of fasted conditions on the bioavailability of VH4004280 Formulation A and alternative, optional formulations, relative to their respective bioavailability under fed conditions in Part 1. The optional Part 3 of the study will assess relative bioavailability of VH4004280 Formulation A to up to 3 alternative formulations, selected from Regimens B, C or D, under fed (lower fat) conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 55years of age.
2. Participants who are overtly healthy.
3. Negative (Severe Acute Respiratory Syndrome Coronavirus 2) SARs-CoV-2 test prior to dosing.
4. Has body mass index (BMI) within the range 19-32 (kg/m2).
5. Participants male at birth must use male condoms, and participants female at birth who are of childbearing potential must be using acceptable forms of birth control.
6. Capable of giving signed informed consent.

Exclusion Criteria:

1. History or presence of disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
2. Abnormal blood pressure.
3. Any malignancy within the past 5 years except certain localized malignancies, or breast cancer within the past 10 years.
4. Has exclusionary psychiatric, hepatic, cardiovascular, gastrointestinal, respiratory, endocrine, neurological, hematological, or renal condition.
5. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
6. Participants with exclusionary electrocardiogram findings.
7. Past or intended use of exclusionary medications or vaccines.
8. Exposure > 4 new investigational products within 12 months, previous participation in this study, or current enrolment or participation in another investigational study.
9. ALT >1.5x upper limit of normal (ULN), total bilirubin >1.5x ULN, and/or estimated serum creatinine clearance <60 mL/min.
10. History of or current infection with hepatitis B or hepatitis C.
11. Positive SARS-CoV-2 test, having signs and symptoms suggestive of COVID-19, or contact with known COVID-19 positive person.
12. Positive HIV antibody test.
13. Participants with positive results for illicit drug use, regular use of drugs of abuse, tobacco or nicotine-containing product use, and/or excessive alcohol use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve from time zero (pre-dose) to infinity time (AUC[0-inf]) of VH4004280 in fed conditions (after a high-fat or lower-fat meal) | From Day 1 to Day 49
Area under the plasma drug concentration - time curve from zero (pre-dose) to the end of the dosing interval at steady state (AUC[0-tlast) of VH4004280 in fed conditions (after a high-fat or lower-fat meal) | From Day 1 to Day 49
Maximum observed plasma drug concentration (Cmax) of VH4004280 in fed conditions(after a high-fat or lower-fat meal) | From Day 1 to Day 49
Time to maximum observed plasma concentration (Tmax) of VH4004280 in fed conditions (after a high-fat or lower-fat meal) | From Day 1 to Day 49

SECONDARY OUTCOMES:
Number of participants with AEs (Adverse Events), by severity | From Day 1 to Day 49
  An AE is any untoward medical occurrence in a participant or clinical investigation participant and can be any sign, symptom, or disease temporally associated with the use of a medicinal product. The severity scale is assessed as following: Grade 1 = mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated. Grade 2 = moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated. Grade 3 = severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated. Grade 4 = potentially life-threatening symptoms causing inability to perform self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.
Number of participants with maximum toxicity grade increase from baseline for liver laboratory parameters | From Day 1 to Day 49
  The assessed laboratory assessments include Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase (ALP), direct bilirubin and total bilirubin, in both fed and fasted conditions.
Change from baseline in liver panel parameters: Total bilirubin and direct bilirubin (micromoles per liter) | From Day 1 to Day 49
Change from baseline in liver panel parameters: ALT, ALP and AST (International units per liter) | From Day 1 to Day 49

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/